CLINICAL TRIAL: NCT07296120
Title: Seroconversion Following RSV Vaccination in Bone Marrow Transplant and CAR-T Patients
Brief Title: RSV Vaccine Response in Stem Cell and CAR-T Therapy Recipients
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Cooper Health System (Other)
Collaborators: The Cooper Foundation (Unknown)
Responsible Party: Principal Investigator, Anil Rengan, Assistant Professor of Medicine, Hematology/Oncology, Cooper University Health Care, Cooper University Health Care
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 25-114
Record Dates: First submitted 2025-12-15; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: CAR-T Cell Therapy; RSV Immunization; Bone Marrow Transplant - Autologous or Allogeneic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vaccine Recipients (Experimental): Patients who will recieve the RSV vaccine
  Interventions: Biological: Respiratory Syncytial Virus Prefusion F Vaccine (RSVpreF)

INTERVENTIONS:
Biological: Respiratory Syncytial Virus Prefusion F Vaccine (RSVpreF) — Patients will receive a single dose of the Respiratory Syncytial Virus Prefusion F Vaccine (RSVpreF) starting at three months post-HSCT or CAR-T therapy.

SUMMARY:
This study evaluates whether the RSV vaccine Abrysvo can produce an antibody response in patients with blood cancers who have previously received a hematopoietic stem cell transplant (HSCT) or CAR-T cell therapy. The vaccine targets the prefusion F (preF) protein of RSV, which is an important component of protective immunity against the virus.

The main goal of the study is to measure the change in antibody levels against the preF protein four weeks after vaccination compared with levels before vaccination. The study will also assess whether participants develop a meaningful immune response, defined as at least a four-fold increase in RSV neutralizing antibody levels four weeks after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosis of hematological malignancy
* Treatment with HSCT or CAR-T therapy
* Must be able to give informed consent
* Must be willing to provide blood samples after HSCT or CAR-T therapy and prior to vaccination
* Must be willing to provide blood samples at four weeks and six months post-vaccination
* Must have an insurance plan that covers the cost of recieving the RSV vaccine.

Exclusion Criteria:

* History of a severe allergic reaction to any component of the RSV vaccine
* Use of intravenous immunoglobulin (IVIG) for hypogammaglobulinemia within the past six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Fold Rise in Antibody Titers and Seroconversion | From the time the patient receives the vaccine to four weeks post-vaccination.
  The primary endpoint is the fold rise in antibody titers against the preF protein at four weeks post-vaccination compared to pre-vaccination (baseline) levels. An additional related objective is to assess whether patients are able to achieve seroconversion. The endpoint for this objective is the proportion of patients with at least a four-fold increase in neutralizing titers from the pre-vaccination baseline at four weeks post-vaccination.

SECONDARY OUTCOMES:
Persistence of Humoral Immune Response | From four weeks post-vaccination to six months post-vaccination
  The secondary objective is to assess whether patients who achieve seroconversion at four weeks post-vaccination retain high levels of neutralizing antibodies at six months post-vaccination. The endpoint for this objective is the fold change in antibody titers against the preF protein at six months post-vaccination compared to four weeks post-vaccination.
COVID-19 and Influenza Immunity | From the collection of baseline antibody titers to the collection of antibody titers at six months post-vaccination against RSV.
  Although vaccination against these pathogens is not part of the study protocol, neutralizing antibody titers for influenza and COVID-19 will be obtained alongside RSV titers as part of a broader titer analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States